CLINICAL TRIAL: NCT03638310
Title: Assessment of Visual Sensitivity, Psychiatric Profile and Quality of Life Following Vestibular Schwannoma Surgery in Patients Prehabituated by Chemical Vestibular Ablation
Brief Title: Role of Psychiatric Profile in Prehabituated Patients After Vestibular Schwannoma Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Balatkova Zuzana, Zuzana Balatkova, M.D., Principal Investigator, Department of otorhinolaryngology and head and neck surgery,1st faculty of medicine Charles university and University hospital Motol, Prague, Head: Prof. Jan Plzak, M.D., Ph.D., Charles University, Czech Republic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13943 FN Motol
Record Dates: First submitted 2018-05-08; First posted 2018-08-20 (Actual); Last update posted 2018-08-20 (Actual); Status verified 2018-08

CONDITIONS: Vestibular Schwannoma; Vestibular Function Disorder
MeSH Terms: conditions — Neuroma, Acoustic; Vestibular Diseases

STUDY DESIGN:
Intervention Model Description: two groups of patients, one group prehabituated by chemical labyrintectomy, the second control group without prehabituation before the surgery
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ITG (intratympanic gentamicin) group (Experimental): Patients who underwent prehabituation by gentamicin prior to surgery for vestibular schwannoma. They underwent intratympanic application of gentamicin and microsurgical removal of vest. schwannoma.
  Interventions: Procedure: intratympanic application of gentamicin; Procedure: microsurgical removal of vestibular schwannoma
- control group (Active Comparator): patients without prehabituation before surgery. They underwent microsurgical removal of vest. schwannoma.
  Interventions: Procedure: microsurgical removal of vestibular schwannoma

INTERVENTIONS:
Procedure: intratympanic application of gentamicin — under local anesthesia is gentamicin instilled through tympanic membrane to tympanic cavity
  Arms: ITG (intratympanic gentamicin) group
Procedure: microsurgical removal of vestibular schwannoma — surgery under general anesthesia

SUMMARY:
The aim of this study is to assess effect of psychiatric profile on visual sensitivity and overall health status in patients who underwent surgery for vestibular schwannoma and were prehabituated by chemical vestibular ablation.

ELIGIBILITY:
Inclusion Criteria:

* T3, T4 vestibular schwannoma
* recorded growth of a tumour
* hearing loss greater than 50% in PTA

Exclusion Criteria:

* T1 vestibular schwannomas
* no growth progression
* normal hearing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
change of optokinetic nystagmus measurement | change of the gain of optokinetic nystagmus among 3 time points is measured: before intervention, 1 week after intervention, 3 months after intervention
  During electronystagmography gain of optokinetic nystagmus is measured before and after the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Zdeněk čada, M.D., Ph.D., Study Chair — Charles university Prague
Locations (1):
- Charles University, Prague, Czechia

IPD SHARING:
Plan to Share IPD: Undecided
It is planned to share the data concerning description of pathology (size of the tumour), outcomes of clinical examination- objective vestibular measures, outcomes of questionnaires (QoL, depression/anxiety scale)

REFERENCES:
- [Background] Cada Z, Balatkova Z, Chovanec M, Cakrt O, Hruba S, Jerabek J, Zverina E, Profant O, Fik Z, Komarc M, Betka J, Kluh J, Cerny R. Vertigo Perception and Quality of Life in Patients after Surgical Treatment of Vestibular Schwannoma with Pretreatment Prehabituation by Chemical Vestibular Ablation. Biomed Res Int. 2016;2016:6767216. doi: 10.1155/2016/6767216. Epub 2016 Dec 8. PMID 28053986
- [Derived] Balatkova Z, Cada Z, Hruba S, Komarc M, Cerny R. Assessment of visual sensation, psychiatric profile and quality of life following vestibular schwannoma surgery in patients prehabituated by chemical vestibular ablation. Biomed Pap Med Fac Univ Palacky Olomouc Czech Repub. 2020 Dec;164(4):444-453. doi: 10.5507/bp.2019.056. Epub 2019 Dec 3. PMID 31796939